CLINICAL TRIAL: NCT00413881
Title: A Prospective Comparison of Alcon LADARVision Wavefront-guided LASIK Enhancement and Conventional LASIK Enhancement for the Correction of Residual Refractive Errors Following LASIK Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRAMC WU # 04-23011
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2008-03

CONDITIONS: Refractive Errors
Keywords: Residual refractive error left over from initial LASIK correction.; Higher Order aberrations measured using a wavefront analyzer.
MeSH Terms: conditions — Refractive Errors

ARMS (2):
- 2 (Active Comparator): Conventional LASIK Enhancement
  Interventions: Procedure: CONVENTIONAL LASIK ENHANCEMENT
- 1 (Experimental): Wavefront guided LASIK Enhancement
  Interventions: Procedure: WAVEFRONT- GUIDED LASIK ENHANCEMENT

INTERVENTIONS:
Procedure: WAVEFRONT- GUIDED LASIK ENHANCEMENT — Laser treatment to correct residual refractive error left over from initial LASIK correction using wavefront guided LADARvision 4000 excimer laser system
  Arms: 1
Procedure: CONVENTIONAL LASIK ENHANCEMENT — Laser treatment to correct residual refractive error left over from initial LASIK correction using LADARvision 4000 excimer laser system.
  Arms: 2

SUMMARY:
The purpose of this study is to conduct a prospective clinical trial to compare conventional and WFG LASIK for enhancements on post-LASIK patients. Differences in safety, efficacy, visual quality, and refractive stability will also be compared during this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any race, and at least 21 years old at the time of the preoperative exam, and have signed an informed consent. The lower age limit of 21 years is intended to ensure documentation of refractive stability.
* At least 6 months from original LASIK surgery.
* Stable refraction with more than 0.75D of spherical equivalent from the desired correction and have less than 1.50D of cylinder in the manifest refraction.
* Both eyes must be within 1.00D spherical equivalent of each other on the manifest refraction test.
* The eye to be treated with wavefront-guided enhancement must have at least a 9.5mm flap.
* Manifest refraction and LADARWave™ refractions must be within 1.00D.
* At least 3 lines potential improvement in UCVA.
* BSCVA of 20/20 or better.
* Good corneal flap and interface.
* Adequate corneal thickness for surgery (residual stromal bed > 280 microns).
* Able and willing to give informed consent.
* Located in the greater Washington DC area for a 12-month period.
* Access to transportation to meet follow-up requirements.

Exclusion Criteria:

* Female subjects who are pregnant, breast-feeding or intend to become pregnant during the study. Pregnancy will be ruled out with a urine pregnancy test.
* Concurrent topical or systemic medications that may impair healing, including corticosteroids, antimetabolites, isotretinoin, amiodarone hydrochloride and/ or sumatripin, as determined by history.
* Medical condition(s), which, in the judgement of the investigator, may impair healing, including but not limited to: collagen vascular disease, autoimmune disease, immunodeficiency diseases, and ocular herpes zoster or simplex (As determined by history).
* Active ophthalmic disease, neovascularization of the cornea within 1mm of the intended ablation zone, or clinically significant lens opacity.
* Evidence of glaucoma or an intraocular pressure greater than 22mm Hg at baseline.
* Evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye.
* Flap irregularity(striae, interface debris, scarring, or epithelium).
* Calculated residual stroma bed less than 280.
* Stable refraction with less than 0.75D of spherical equivalent from the desired correction and more than 1.5D of cylinder in the manifest refraction.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-07; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
1.Safety 2. Efficacy 3. Refractive stability | one year after enhancement

CONTACTS AND LOCATIONS:
Overall Officials: RICHARD STUTZMAN, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Center For Refractive Surgery, Washington D.C., District of Columbia, United States